CLINICAL TRIAL: NCT04063813
Title: Parameters of Exercise to Prevent Osteoporosis
Acronym: OSTEOPOROSISEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Wisconsin, La Crosse (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dr. Katarina Borer, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00007202
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: Five parallel groups, matched for age and BMI, where exercise was applied at 6o uphill or 6o downhill either as one 40-min morning bout or as two 20-min half bouts distributed 7 h apart. A sedentary group served as a control for the four exercise groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 40 minute up trial (Experimental): Subjects were subjected to 40 minutes of treadmill exercise at a 6 degree incline and at 75% of maximal effort between 8:00 and 8:40 am. Isocaloric meals were provided at 7:00, 13:00. and 19:00 h.
  Interventions: Behavioral: Experimental: 40 minute up trial
- 40 minute down trial (Experimental): Subjects were subjected to 40 minutes of treadmill exercise at a 6 degree decline and at 45% of maximal effort between 8:00 and 8:40 am. Isocaloric meals were provided at 7:00, 13:00. and 19:00 h.
  Interventions: Behavioral: Experimental: 40 minute down trial
- Two 20 minute up trials (Experimental): Subjects were subjected to two 20 minutes of treadmill exercise separated by 7 h at a 6 degree incline and at 75% of maximal effort, the first one between 8:00 and 8:40 am and the second one between 15:00 and 15:20 h..Isocaloric meals were provided at 7:00, 13:00. and 19:00 h.
  Interventions: Behavioral: Experimental: Two 20 minute up trials
- Two 20 min down trials (Experimental): Subjects were subjected to two 20 minutes of treadmill exercise separated by 7 h at a 6 degree incline and at 45% of maximal effort , the first one between 8:00 and 8:40 am and the second one between 15:00 and 15:20 h. Isocaloric meals were provided at 7:00, 13:00. and 19:00 h.
  Interventions: Behavioral: Experimental: Two 20 min down trials
- Sedentary trial (Active Comparator): No exercise day with isocaloric meals provided at 7:00, 13:00. and 19:00 h.
  Interventions: Behavioral: Active Comparator: Sedentary trial

INTERVENTIONS:
Behavioral: Experimental: 40 minute up trial
  Other Names: 40 minutes of uphill exercise divided into two 20-minute trials separated by 7 h
  Arms: 40 minute up trial
Behavioral: Experimental: 40 minute down trial
  Other Names: 40 minutes of downhill exercise divided into two 20-minute trials separated by 7 h
  Arms: 40 minute down trial
Behavioral: Experimental: Two 20 minute up trials
  Other Names: 40 minutes of uphill exercise separated in two 20-min bouts 7 h apart
  Arms: Two 20 minute up trials
Behavioral: Experimental: Two 20 min down trials
  Other Names: 40 minutes of uphill exercise separated in two 20-min bouts 7 h apart
  Arms: Two 20 min down trials
Behavioral: Active Comparator: Sedentary trial
  Other Names: A control no-exercise trial
  Arms: Sedentary trial

SUMMARY:
The principal goal of this study is to determine parameters of walking in terms of peak mechanical vertical force, bout duration, and bout spacing that can preserve or increase bone mineral density (BMD) in postmenopausal women. Release of pulses of parathyroid hormone (PTH), growth hormone (GH), and of markers of bone resorption and bone formation will be used as indicators of the osteogenic effects of a short exposure to exercise. When secreted in pulsatile fashion, GH stimulates osteoblast proliferation, particularly in cortical bone (27, 28). Like GH, the pattern of PTH secretion determines the nature of its effect on bone. When it is secreted in pulsatile manner, PTH contributes to bone formation through activation of bone lining cells, differentiation of osteoprogenitor cells, and suppression of bone cell apoptosis .

DETAILED DESCRIPTION:
A. Hypotheses and specific aims:

Specific aim 1. Measure plasma concentrations of anabolic hormones (parathyroid hormone (PTH) and growth hormone (GH), at sufficient frequency to define the area under the curve (AUC), and of markers of bone formation (osteocalcin, carboxyterminal propeptide of type 1 procollagen (CICP), and bone-specific alkaline phosphatase (ALKP)), and markers of bone resorption (immunoreactive carboxyterminal telopeptide of type I collagen (CTX)) after 40-minutes of treadmill exercise at the relative intensity of 125% of the ventilatory threshold (VT) corresponding to about 1.78 m/sec (4 miles/h), and two intensities of mechanical loading (724, and 1411 N), in healthy postmenopausal women.

Hypothesis 1. Bone formation, as assessed by increases in markers of bone formation and decreases in markers of bone resorption, will be higher in response to dynamic exercise at a level of mechanical loading that produces increased secretion of PTH and GH than to exercise at other loading intensities.

Specific aim 2. Measure plasma concentrations of anabolic hormones), at sufficient frequency to define the area under the curve (AUC), and of markers of bone formation as in specific aim 1, after two 20-minutes of treadmill exercise, separated by 7 h, at the relative intensity of 125% of the ventilatory threshold (VT) corresponding to about 1.78 m/sec (4 mi/h), and two intensities of mechanical loading (724, and 1411 N), in healthy postmenopausal women.

Hypothesis 2. A 7-hour interval separating the two bouts of exercise will have greater bone anabolic effect than the equivalent volume and intensity of exercise performed in a single bout.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 65 years if naturally post-menopausal, or age 47 if surgically postmenopausal
* Dual energy X-ray absorptiometry (DEXA) Z score above -1
* No endocrine or metabolic disease requiring medication except for hormonally corrected hypothyroidism
* No musculo-skeletal disabilities that would preclude treadmill walking
* Normal electrocardiogram (EKG) and heart health history
* BMI between 24 and 30
* Hematocrit above 32 %
* No hormone replacement therapy (HRT)
* Personal health provider's Release Letter

Exclusion Criteria:

* Age and BMI outside of the specified range
* Z score below -1
* Medication for presence of metabolic or endocrine disease
* Musculo-skeletal disabilities that would preclude treadmill walking
* Abnormal electrocardiogram (EKG) and heart health history
* Hematocrit below 32%
* Hormone replacement therapy
* Failure to conform to study protocol

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 40 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2010-08-19 (Actual); Study Completion 2010-08-19 (Actual)

PRIMARY OUTCOMES:
Ground reaction forces | During last 5 minutes of treadmill walking
  Sum of pressures on mechanosensitive Novel-Pedar shoe insoles
Serum osteocalcin | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of osteocalcin measured in serum samples
Serum CICP (c-terminal propeptide of type 1 collagen | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of CICP measured in serum samples
Serum CTX (c-terminal telopeptide of type 1 collagen | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of CTX measured in serum samples

SECONDARY OUTCOMES:
Relative aerobic capacity | 1 day (measured throughout treadmill exercise bouts)
  Percent of maximal aerobic capacity used during uphill and downhill exercise
Serum insulin | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of insulin measured in serum samples
Serum cortisol | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of cortisol measured in serum samples
Serum GH (growth hormone) | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of GH measured in serum samples
serum PTH (parathyroid hormone) | Hourly blood draws between 8:00 and 22:00 hours
  Concentration of PTH measured in serum samples

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Clinical Research Unit United States, Ann Arbor, Michigan, United States